CLINICAL TRIAL: NCT06412042
Title: Prospective, Placebo-Controlled, Randomized Double-Blind Clinical Study on the Intervention of Animal-Derived Probiotic in Infant Growth and Development, Allergy Incidence, and Immune Function
Brief Title: Probiotic in Infant Growth, Allergy and Immunity Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WK2024006
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Infant ALL

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic BLa80 (Experimental): Participants receive one sachet per day containing probiotic BLa80 and maltodextrin (Day 0 to Day 84).
  Interventions: Dietary Supplement: Probiotic BLa80
- Maltodextrin (Placebo Comparator): Participants receive one sachet per day containing maltodextrin only, serving as the placebo (Day 0 to Day 84).
  Interventions: Other: Placebo Maltodextrin
- Blank (No Intervention): Participants in this arm will not receive any intervention or placebo.

INTERVENTIONS:
Dietary Supplement: Probiotic BLa80 — Collect baby fecal samples, test for 16S rRNA, and analyze changes in the gut microbiota before and after supplementation.
  Arms: Probiotic BLa80
Other: Placebo Maltodextrin — Collect baby fecal samples, test for 16S rRNA, and analyze changes in the gut microbiota before and after supplementation.
  Arms: Maltodextrin

SUMMARY:
To evaluate the intervention effects of Bifidobacterium animalis subsp. lactis strain BLa80 in promoting growth and development (including gut microbiota and physical growth and development) of healthy infants and young children across different age groups, enhancing immune function, improving allergy incidence, and analyzing the safety of BLa80 in relation to infant growth and development, allergy incidence, and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants and young children born at 37 to 42 weeks of gestation through both artificial breastfeeding, with a birth weight greater than or equal to 2500 g and less than 4000 g, regardless of gender
2. Infants and young children whose mothers do not have diagnosed metabolic disorders such as diabetes and are not afflicted with communicable diseases such as hepatitis B or HIV
3. Enrollment will be stratified into three age groups: 0-6 months, 6-12 months, and 12-36 months
4. Consent from parents or primary caregivers of infants and young children to collect faecal samples during the study
5. No clinically diagnosed allergic diseases at the time of enrolment (including but not limited to eczema, asthma, allergic colitis, allergic rhinitis, pollen allergies, etc.)
6. Infants and young children with a medical record established at local maternal and child health care hospital's paediatrics department, undergoing regular check-ups, and following feeding advice and guidance from pediatricians
7. Assurance from family members or primary caregivers not to administer additional probiotic products (including formula milk containing probiotics) to infants and young children during the intervention period.

Exclusion Criteria:

* Healthy infants and young children aged 0-6 months:

  1. Infants with a history of asphyxia at birth or a history of NICU hospitalization
  2. Infants born with congenital defects or abnormalities
  3. Infants whose mother had pregnancy-related conditions such as gestational hypertension, pre-eclampsia or eclampsia, gestational diabetes, cholestasis of pregnancy, or other high-risk obstetric factors, as well as a history of alcohol or drug abuse during pregnancy
  4. Infants who have used antibiotics within 2 weeks prior to enrollment
  5. Infants who have had specific diseases affecting growth and development within 1 month prior to enrollment (e.g., pneumonia, severe diarrhea, severe constipation, severe cow's milk protein allergy, malnutrition, gastrointestinal surgery, severe congenital heart disease, epilepsy, cerebral palsy, developmental delay, confirmed genetic metabolic disorders, chromosomal disorders, genetic diseases, etc.)
  6. Infants with severe primary diseases affecting other important organs or systems such as the heart, liver, kidney, hematopoietic system, etc.
  7. Infants who have used investigational drugs or participated in other clinical studies before screening
  8. Infants who have consumed probiotic products within 1 month prior to enrollment (calculated from birth to enrollment for infants aged <1 month)
  9. Infants who have used immunosuppressive drugs (such as glucocorticoids, immunosuppressants) before enrollment
  10. Infants with known allergies to the ingredients of probiotic products
  11. Children who require hospitalization for treatment due to malnutrition
  12. Other reasons that researchers consider as unsuitable for participation in the clinical trial, such as those that could affect efficacy evaluation or individuals with poor compliance

Infants and young children aged 6-12 months with good health

1. Infants who have used antibiotics within 2 weeks prior to enrollment
2. Infants who have had specific diseases affecting growth and development within the 1 month prior to enrollment (Infants who have had specific diseases affecting growth and development within 1 month prior to enrollment (e.g., pneumonia, severe diarrhea, severe constipation, severe cow's milk protein allergy, malnutrition, gastrointestinal surgery, severe congenital heart disease, epilepsy, cerebral palsy, developmental delay, confirmed genetic metabolic disorders, chromosomal disorders, genetic diseases, etc.)
3. Infants with severe primary diseases affecting other important organs or systems such as the heart, liver, kidney, hematopoietic system, etc.
4. Infants who have used investigational drugs or participated in other clinical studies within 3 months prior to screening
5. Infants who have consumed probiotic products within 1 month prior to enrollment
6. Infants who have used immunosuppressive drugs (such as glucocorticoids, immunosuppressants) before enrollment
7. Infants with known allergies to the ingredients of probiotic products
8. Children who require hospitalization for treatment due to malnutrition
9. Other reasons that researchers consider as unsuitable for participation in the clinical trial, such as those that could affect efficacy evaluation or individuals with poor compliance

Infants and young children aged 12-36 months with good health

1. Infants who have used antibiotics within 2 weeks prior to enrollment
2. Infants who have had specific diseases affecting growth and development within the 1 month prior to enrollment, such as pneumonia, severe diarrhea, severe constipation, severe cow's milk protein allergy, malnutrition, gastrointestinal surgery, severe congenital heart disease, epilepsy, cerebral palsy, developmental delay, confirmed genetic metabolic disorders, chromosomal disorders, genetic diseases, etc.
3. Infants with severe primary diseases affecting other important organs or systems such as the heart, liver, kidney, hematopoietic system, etc.
4. Infants who have used investigational drugs or participated in other clinical studies within 3 months prior to screening
5. Infants who have consumed probiotic products within 1 month prior to enrollment
6. Infants who have used immunosuppressive drugs (such as glucocorticoids, immunosuppressants) before enrollment
7. Infants with known allergies to the ingredients of probiotic products
8. Children who require hospitalization for treatment due to malnutrition
9. Other reasons that researchers consider as unsuitable for participation in the clinical trial, such as those that could affect efficacy evaluation or individuals with poor compliance

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota | 84 days
  Collect patient fecal samples, test for 16S rRNA.

CONTACTS AND LOCATIONS:
Overall Officials: Natalina Soesilawati, Dr., Principal Investigator — Karya Medika II Hospital
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, Jakarta 10430, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided